CLINICAL TRIAL: NCT02608333
Title: Impact of Early Intervention on the Global Development of Children With Autism Spectrum Disorder in a European French-speaking Population Dr Marie-Maude GEOFFRAY Le Vinatier Hospital
Brief Title: Efficiency of Early Intervention for Autism Spectrum Disorder
Acronym: IDEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Collaborators: University Hospital, Strasbourg, France (Other); Versailles Hospital (Other); Centre hospitalier Saint Jean de Dieu - ARHM (Other); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-A00124-45
Record Dates: First submitted 2015-05-11; First posted 2015-11-18 (Estimated); Last update posted 2021-07-09 (Actual); Status verified 2021-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Early intervention; ESDM; behavioral and developmental intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Behavior | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ESDM-12 (Experimental): ESDM -12 : 60 children will receive 12 hours a week of ESDM ( Early Start Denver Model)intervention delivered by trained therapists during 2 years.ESDM is a comprehensive relational, developmental and behavioral intervention.It's described in a manual for Professional and parents.
  Interventions: Behavioral: ESDM-12
- Control group (Active Comparator): control group: 120 children will receive heterogeneous 'as-usual' intervention proposed by professionals and public services over the same period
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: ESDM-12 — ESDM is a comprehensive relational, developmental and behavioral intervention. It's described in a manual for professional (Rogers et al, 2010).
  Children receive ESDM 12H per week by trained therapist. Therapist work in collaboration with parents (at home) and preschool or nursery.
  Other Names: Early Start Denver Model 12 hours per week
  Arms: ESDM-12
Behavioral: control group — heteregenous "as usual "community intervention
  Arms: Control group

SUMMARY:
Intervention for autism spectrum disorder (ASD) in European French-speaking countries is often heterogeneous and poorly evaluated. Six French-speaking early intervention units for children with ASD following the Early Start Denver Model (ESDM) have been created since 2011 with the common aim to evaluate effectiveness and cost-efficiency of the ESDM applied to the European French-speaking public health system. In those units, Children receive ESDM at minimum 12H per week by trained therapist. Therapist work in collaboration with parents (at home) and preschool or nursery.

The first aim of the investigators study is to evaluate the effectiveness of ESDM intervention 12 hours per week during 2 years on the global development of children with ASD compared to the interventions commonly available in the community.

DETAILED DESCRIPTION:
This is a multicenter (4 centers in France, 1 center in Switzerland and 1 center in Belgium), randomized, controlled, single blind trial using a modified Zelen design .It concerns children with ASD aged 18 to 36 months without severe neurological or physical disorder and living in the proximity of one the early intervention units. After diagnostic, Children will be included in a longitudinal cohort with the consent of the parents. Sixty children will be drawn lots among 180 children of the cohort and will be included in a ESDM intervention with the consent of the parents. Two groups will be compared: an experimental group of 60 children receiving 12 hours a week of ESDM intervention delivered by trained therapists during 2 years and a control group of 120 children receiving typical heterogeneous 'as-usual' intervention proposed by professionals and public services over the same period. Global developmental profiles of all the children will be measured at different time points over the two years through standardized tests such as the Mullen Scale of Early Learning (MSEL), the ADOS-2 and the Vineland Adaptive Behavior Scale. Cost of each intervention will be calculated.

The primary outcome is global development of the child, measured by the developmental quotient with the Mullen after 24 months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children 15 months to 36 months
* Children with autism spectrum disorder (according to international criteria and standardized tests)
* Children at a DQ of 30 at least at the MSEL
* Family domiciled within 40 minutes of a early intervention unit (investigator center for the study)

Exclusion Criteria:

* Severe neurological or physical disorder identified not allowing intensive care
* Unavailability of the family for regular monitoring of the child by the investigator center
* Rett Syndrom

Ages: 15 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Developmental quotient at the Mullen Scale of Early Learning | Change from baseline in developmental quotient at 24 months follow-up
  This criterion will be assessed with the Mullen scale of Early Learning (Mullen, 1995) by a psychologist blind of intervention group of the child:

SECONDARY OUTCOMES:
Severity of autism symptoms is measured with ADOS 2 | Change from baseline in severity score of autism symptoms at 24 months follow-up
  severity of autism symptoms is measured with ADOS 2 ( Autism Diagnostic observation Schedule 2)
Adaptive behavior score is measured by the composite score of Vineland adaptative behavior scale 2 | Change from baseline in adaptative behavior at 24 months follow-up
  Adaptative behavior score is measured by the composite score of Vineland adaptative behavior scale 2
Productive language level assessed with a standardized French productive language developmental scale | change from baseline in number of words at 24 months follow-up (T2)
  This criterion will be assessed with a standardized French productive language developmental scale (DLPF "Development du language de production" in French language) filled by parents
Costs associated with interventions | at 24 months follow-up (T2)
  Healthcare, social and personal resources devoted to child care throughout the study will be measured to evaluate the direct and indirect costs associated with intervention. Assessment will take place
Developement of communication and symbolic behavior | At baseline (inclusion ° T0), at 12 months follow-up (T1), and at 24 months follow-up
  Total score of Communication and Symbolic Behaviour Scale Developmental Profil CSBS-DP questionnaire for caregivers (Wetherby et al, 2002)
Parent child naturalistic interaction during play | At baseline (inclusion ° T0), at 12 months follow-up (T1), and at 24 months follow-up (T2)
  Dyadic Communication Measure for Autism (DCMA)(Green et al, 2010; Pickles, 2015) will be used and score of parent's communication synchrony, child initiation, and shared attention will be assessed
Sensorial profil | At baseline (inclusion ° T0), at 12 months follow-up (T1), and at 24 months follow-up (T2)
  Sensorial profil of Dunn
Change at the Brief Observation of Social Communication Change (BOSCC) | At baseline (inclusion ° T0), at 12 months follow-up (T1), and at 24 months follow-up
  The total score of Brief Observation of Social Communication Change

CONTACTS AND LOCATIONS:
Overall Officials: GEOFFRAY MARIE-MAUDE, DR, Principal Investigator — CH LE VINATIER
Locations (1):
- Hopital Vinatier, Bron, AURA, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Geoffray MM, Oreve MJ, Jurek L, Sonie S, Schroder C, Delvenne V, Manificat S, Touzet S, Agathe J, Mengarelli F, Natacha G, Petit N, Speranza M, Bahrami S, Bouveret L, Dochez SL, Auphan P, Zelmar A, Falissard B, Carlier S, Nourredine M, Denis A, Febvey-Combes O. Early Start Denver Model effectiveness in young autistic children: a large multicentric randomised controlled trial in two European countries. BMJ Ment Health. 2025 Jun 5;28(1):e301424. doi: 10.1136/bmjment-2024-301424. PMID 40473417
- [Derived] Touzet S, Occelli P, Schroder C, Manificat S, Gicquel L, Stanciu R, Schaer M, Oreve MJ, Speranza M, Denis A, Zelmar A, Falissard B, Georgieff N, Bahrami S, Geoffray MM; IDEA Study Group. Impact of the Early Start Denver Model on the cognitive level of children with autism spectrum disorder: study protocol for a randomised controlled trial using a two-stage Zelen design. BMJ Open. 2017 Mar 27;7(3):e014730. doi: 10.1136/bmjopen-2016-014730. PMID 28348195